CLINICAL TRIAL: NCT03801590
Title: Safety and Efficacy Of Corneal Collagen Crosslinking (CXL) In Infectious Keratitis
Brief Title: Crosslinking in Infectious Keratitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Asem, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: infectious keratitis
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Infectious Keratitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXL on patients with infectious keratitis (Experimental): the procedure of cross linking(CXL) :combined riboflavin-ultraviolet type A rays (UVA) collagen cross-linking. Radiant energy was 3 milliwatts/cm2 for a 30-minute exposure irradiation of the cornea will be carried out on twenty patients with infectious keratitis .
  Interventions: Device: Crosslinking with Riboflavin and UV-A

INTERVENTIONS:
Device: Crosslinking with Riboflavin and UV-A — the procedure of cross linking(CXL) :combined riboflavin-ultraviolet type A rays (UVA) collagen cross-linking. Radiant energy was 3 milliwatts/cm2 for a 30-minute exposure irradiation of the cornea.

SUMMARY:
Microbial keratitis is an infection of the cornea that is associated with risk of permanent visual impairment.

It can be caused by bacteria, virus, fungus, protozoa and parasites. The common risk factors for infectious keratitis include ocular trauma, contact lens wear, recent ocular surgery, preexisting ocular surface disease, dry eyes, lid deformity, corneal sensation impairment, chronic use of topical steroids and systemic immunosuppression .

DETAILED DESCRIPTION:
The spectrum of bacterial keratitis can also be influenced by geographic and climatic factors.

The treatment usually consist of Topical administered antibiotics .the emergence of multidrug-resistant bacteria is a concern that might complicate the treatment and cure of infectious keratitis.

Collagen cross linking (CXL) using ultraviolet-A (UV-A) and riboflavin in a treatment that was developed to increase the biochemical strength of the cornea The procedure is based on using riboflavin as a photosensitizer, which generates reactive oxygen species when activated by UV-A at 365 or370 nm.

The standard technique (epi-off) also called Dresden Protocol includes removal of the epithelium in order to expose the underlying stroma to riboflavin, which is otherwise incompletely absorbed by the epithelium because of tight junctions. The area of corneal epithelium removed has a diameter of 6.0 to 8.5 mm. A crosslinking procedure without epithelial removal could also be performed (epi-on). It would likely be less painful compared to the standard procedure.

The crosslinking process generates reactive oxygen species that can damage the cell walls of pathogens. CXL induces formation of new covalent bonds thereby rendering the corneal stroma biomechanically stronger and more resistant to enzymatic digestion . This can potentially limit the spread of infection. Furthermore, CXL-induced apoptosis could contribute to the reduction of inflammatory response during corneal infection .

ELIGIBILITY:
Inclusion Criteria:

* Patients with proved bacterial, fungal, acanthamoeba microbial keratitis .
* Patient willing to comply with all study procedures .

Exclusion Criteria:

* Severe corneal scarring or opacification .
* Patients with viral infectious keratitis
* Prior herpetic infections .
* Patients with any coexisting ocular pathology,ocular surface disease .
* Patients with Autoimmune disease.
* Pregnant women .
* Corneal Thickness of less than 400 microns .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine the duration for corneal ulcer healing | one year
  By follow up with photography before crosslinking and one week after performing cxl.

REFERENCES:
- [Background] Green M, Apel A, Stapleton F. Risk factors and causative organisms in microbial keratitis. Cornea. 2008 Jan;27(1):22-7. doi: 10.1097/ICO.0b013e318156caf2. PMID 18245962
- [Background] Jankov Ii MR, Jovanovic V, Nikolic L, Lake JC, Kymionis G, Coskunseven E. Corneal collagen cross-linking. Middle East Afr J Ophthalmol. 2010 Jan;17(1):21-7. doi: 10.4103/0974-9233.61213. PMID 20543933